CLINICAL TRIAL: NCT06000605
Title: Does Cerebral Substrate Switching Underlie the Beneficial Brain Adaptations of Fasting and Exercise?
Brief Title: Brain Substrate Switch to Ketones and Lactate
Acronym: BSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Collaborators: University of Otago (Other)
Responsible Party: Principal Investigator, Phil Ainslie, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Brain_substrate_switch
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Metabolic Diseases; Aging Problems
Keywords: brain; BDNF; metabolism; ketones; lactate
MeSH Terms: conditions — Metabolic Diseases; Ketosis

STUDY DESIGN:
Intervention Model Description: Participants will complete both arms: 1) fasted and 2) fed.
Who Masked: Investigator
Masking Description: The participant will not be blinded because they must consciously adhere to study requirements, i.e., fasting for 3 days. The investigators will be blinded to the fasting and fed conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fed (Active Comparator): Exercise and passive infusions of ketones and lactate in the fed state. Participants will be fed a small meal in the middle of the protocol, also.
  Interventions: Other: Fed
- Fasted (Experimental): Exercise and passive infusions of ketones and lactate in the fasted state. Participants will be required to fast for 72 hours prior to arriving to the lab for this testing arm.
  Interventions: Other: Fasted

INTERVENTIONS:
Other: Fed — Participants will eat a light meal prior to testing and be fed a light meal during testing.
  Arms: Fed
Other: Fasted — Participants will completely abstain from calories for 72 hours prior to testing and not receive any calories during testing.
  Arms: Fasted

SUMMARY:
The brain is constantly active and energetically expensive, making up a quarter of the body's energy budget despite occupying only 2% of its mass. To fuel this incessant activity, the brain relies on glucose, which accommodates 99% of its metabolic needs. In most cases, glucose is the ideal fuel since it is in constant surplus owing to 24-hr access to sugar-rich food. However, the brain is metabolically flexible and capable of metabolizing alternative fuels when glucose is scarce, or, decreasing rapidly. For example, during fasting when glucose stores are dwindling, ketone bodies can supplement the brain's metabolic needs. During intense exercise, when glucose stores are being rapidly depleted, lactate - a byproduct of this glucose turnover - similarly acts as an alternative fuel for the brain. In healthy individuals, exploiting this 'brain metabolic flexibility' may be beneficial in protecting the brain from aging.

The main question is: Does the brain substrate switch that occurs during fasting and high-intensity exercise underlie the beneficial effects on the brain?

Young, healthy participants will fast for 3 days and complete high-intensity cycling exercise, each of which will induce a brain substrate switch. Participants will also be passively infused with ketones (to simulate fasting) and lactate (to simulate high-intensity exercise) in the fed and rested state. In doing so, the investigators will isolate the brain substrate switch from the broader, pluripotent stressors that encompass fasting and exercise.

The main outcome variables are the brain biomarkers: brain-derived neurotrophic factor (BDNF) and secreted amyloid beta precursor protein (sAPPA).

DETAILED DESCRIPTION:
Objectives:

Primary:

• To determine if brain ketone and lactate metabolism cause the beneficial neurotrophic responses associated with fasting and exercise, respectively.

Secondary:

• To determine if fasting and exercise improve the brain's uptake of glucose, ketones and lactate.

Endpoints:

Primary:

* Brain-derived neurotrophic factor (BDNF)
* Secreted amyloid-beta precursor protein-alpha (sAPPA)

Secondary:

* Brain glucose extraction
* Brain ketone extraction
* Brain lactate extraction
* Increased brain glucose extraction in response to intra-nasal insulin administration

Hypothesis:

1. Fasting and high-intensity exercise will increase the brain's release of BDNF and sAPPA, and these responses will be the same when ketones and lactate are passively infused into circulation in the fed and rested state.
2. Fasting will increase brain ketone metabolism beyond that achieved when ketones are passively infused into circulation in the fed state.
3. High-intensity exercise will increase brain lactate metabolism beyond that achieved when lactate is passively infused into circulation in the rested state.
4. High-intensity exercise will improve the brain's insulin sensitivity to glucose, as shown by increase brain glucose uptake in response to intra-nasal insulin.

Design

This will be a repeated-measures cross-over design with participants completing two conditions separated by 4-6 weeks:

1. Fed exercise and passive infusions of lactate and ketones
2. 72-hr fasted exercise and passive infusions of lactate and ketones

On both visits, participants will be instrumented with arterial (radial) and venous (internal jugular) catheters to quantify cerebral oxidative and substrate (glucose, ketones, lactate) metabolism in response to: 1) fasting, 2) 6 minutes of high-intensity exercise, 3) a passive graded infusion of ketones (to mimic fasting); and 4) a passive graded infusion of lactate (to mimic exercise). Brain insulin sensitivity to glucose will be quantified in the fed and fasted states before and after exercise by a one-time dose of intranasal insulin. In the fed and fasted states at rest, a cerebrospinal fluid sample will be collected from the lumbar spine to quantify metabolomics and the production and release of neurotrophic factors (BDNF and sAPPa) from the brain.

Trial Sites All testing will take place in the ARTs Building (Room 184) in the Centre for Heart, Lung and Vascular Health research laboratory in Kelowna, British Columbia, Canada.

Participants Sample size The investigators will collect data in 12 subjects with both sexes included. A sample size calculation (power >0.8, significance < 0.05) based on our preliminary data indicates 8 participants are required; the investigators will aim to recruit 12 volunteers of both sexes to better represent the population, not to investigate sex differences. Written, informed consent will be obtained from participants. The investigators anticipate a dropout rate of <5%.

Inclusion criteria

* Aged 19 - 40 years old
* Regularly physically active, as determined via questionnaires

Exclusion criteria

* Current smokers
* Acute bronchial asthma, chronic obstructive airway or status asthmaticus
* Obese (body mass index greater than 30 kg m-2)
* Requiring daily prescription medications that may affect responses to exercise, e.g., anti-hypertensives, anti-arrhythmogenics, inhalers
* History of disease/dysfunction that could cause complication with exercise, e.g. cardiovascular, respiratory, neurological or musculoskeletal diseases
* Irregular or absent menstrual cycle (females)
* Pregnant or may suspect pregnancy, or post-menopausal (females)
* Any unexpected adverse responses to pre-experimental exercise tests
* Any contraindication to a lumbar subarachnoid access

Screening/Baseline Evaluation

The above inclusion and exclusion criteria will be examined via a health screening questionnaire and a clinical screening performed by a physician. This screening will include:

* Resting blood pressure,
* 12-lead electrocardiogram,
* Cardiopulmonary exercise testing,
* Fasting blood glucose.

Discontinuation criteria

• Any adverse response to invasive procedures, i.e., catheterization and cerebrospinal fluid sampling (please see Risks below)

In addition to the above and as per UBC Clinical Research Ethics Board guidelines, all research participants are able to withdraw from the study at any time and without reason.

Experimental procedures

Participants will visit the lab on two occasions. Details of the experimental visits are outlined below:

1. Fed exercise and passive infusions of lactate and ketones

   Participants will arrive to the lab 1 hr after eating a light meal of their choice. Participants will lie on a bed and will be instrumented with indwelling radial artery and internal jugular vein catheters. One hour after catheterizations, cerebral blood flow will be measured non-invasively by Duplex ultrasound of the internal carotid and vertebral arteries. Blood samples will be collected from the arterial and venous circulations for resting measures of brain oxidative and substrate (glucose, ketones and lactate) metabolism. A single cerebrospinal fluid sample will be collected from the lumbar spine between L4 and L5. This procedure will be performed by a highly trained physician who uses these techniques routinely for patient care on a near daily basis. Thereafter, the primary ketone, beta-hydroxybutyrate (Bhb), will be infused via an antecubital (arm) vein in a stepwise manner to induce circulating concentrations of 1, 3 and 5 mmol/L. Following a complete recovery, i.e., Bhb concentration return to resting values, intravenous lactate will be infused in a stepwise manner to induce circulating concentrations of 5, 10 and 15 mmol/L. Following a complete recovery of blood lactate levels, an intravenous combined infusion (Bhb and lactate) will be administered to induce circulating concentrations of 3 and 10 mmol/L, respectively. Participants will then be given a light standardized meal and 1 hour to rest and digest. Lastly, participants will self-administer a single-dose of intranasal insulin before and after completing 6-minutes of high-intensity cycling intervals. After the final dose of intranasal insulin, participants will be de-instrumented marking the end of the visit. The total time for this visit is estimated to be 3-4 hours.
2. 72-hr fasted exercise and passive infusions of lactate and ketones

This visit is identical to condition 1, except that participants will arrive at the lab 72 hr fasted and will not be provided with a light meal until completion of all experimental procedures. Prior to initiating the fast, participants will be equipped with a continuous glucose monitor so that the researchers can track their blood glucose during the fast. As such, the total time for this visit is also estimated to be 3-4 hours.

High-intensity exercise protocol. Participants will complete six 40-s bouts of cycling at a work rate that elicits 100% maximal aerobic power (V̇O2max) followed by 20 s of active recovery at 25% VO2max. The investigators have shown this exercise bout to increase lactate >5-fold in both the fed and fasted state.

Randomization of conditions. The order of conditions, i.e., fed or fasted, will be randomized. It is impossible to blind the participants to the fed and fasted conditions since fasting requires abstaining for eating prior to visiting the lab. Researchers will not be blinded because they will be monitoring the subjects while they are fasting prior to visiting the lab.

ELIGIBILITY:
Inclusion Criteria:

* Regularly physically active, as determined via questionnaires

Exclusion Criteria:

* Current smokers
* Acute bronchial asthma, chronic obstructive airway or status asthmaticus
* Obese (body mass index greater than 30 kg m-2)
* Requiring daily prescription medications that may affect responses to exercise, e.g., anti-hypertensives, anti-arrhythmogenics, inhalers
* History of disease/dysfunction that could cause complication with exercise, e.g. cardiovascular, respiratory, neurological or musculoskeletal diseases
* Irregular or absent menstrual cycle (females)
* Pregnant or may suspect pregnancy, or post-menopausal (females)
* Any unexpected adverse responses to pre-experimental exercise tests
* Any contraindication to a lumbar subarachnoid access

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Brain-derived neurotrophic factor, secreted amyloid beta precursor protein | Data collected at rest, during graded infusions of lactate and ketones, pre- and post- 6 minutes of high-intensity cycling exercise
  Biomarker to index neuroplasticity and resilience

SECONDARY OUTCOMES:
Brain substrate metabolism | Data collected at rest, during graded infusions of lactate and ketones, pre- and post- 6 minutes of high-intensity cycling exercise
  The brain's turnover of glucose, beta-hydroxybutyrate (ketone body) and lactate

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia - Okanagan Campus, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
No personal data will be made available publicly or to other researchers.